CLINICAL TRIAL: NCT00006267
Title: A Phase II Evaluation Of 9-Nitro-Camptothecin In The Third-Line Treatment Of Recurrent Ovarian Or Primary Peritoneal Cancer
Brief Title: Nitrocamptothecin in Treating Patients With Recurrent or Metastatic Ovarian Epithelial or Primary Peritoneal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Never activated.
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000068210; GOG-0186B
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2004-05

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — rubitecan

INTERVENTIONS:
Drug: rubitecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of nitrocamptothecin in treating patients who have recurrent or metastatic ovarian epithelial or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of nitrocamptothecin in patients with recurrent or metastatic ovarian epithelial or primary peritoneal cancer.
* Determine the nature and degree of toxicity of this regimen in these patients.

OUTLINE: Patients receive oral nitrocamptothecin on days 1-5. Treatment continues every 7 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 2 weeks, then every 3 months for 2 years, and then every 6 months for 3 years.

PROJECTED ACCRUAL: Approximately 19-51 patients will be accrued for this study within 22 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or metastatic ovarian epithelial or primary peritoneal cancer
* Measurable disease

  * Ascites and pleural effusions are not considered measurable
  * Sonography allowed if bidimensionally measurable
* Must not be eligible for higher priority GOG protocol

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Granulocyte count at least 1,500/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT and alkaline phosphatase no greater than 3 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* No other prior or concurrent invasive malignancy in the past 5 years except nonmelanoma skin cancer
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least but no more than 2 prior chemotherapy regimens containing carboplatin, cisplatin, or another organoplatinum compound combined with paclitaxel
* Second line therapy may include any agents except topoisomerase I inhibitors (i.e., topotecan)
* No prior nitrocamptothecin or topoisomerase I inhibitors
* At least 3 weeks since prior chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered

Surgery:

* At least 3 weeks since prior surgery and recovered

Other:

* No prior cancer therapy that contraindicates this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward C. Grendys, MD, Study Chair — Robert H. Lurie Cancer Center